CLINICAL TRIAL: NCT01443624
Title: Evaluation of Oxidative Stress Induced by Iron Injection in Healthy Volunteers Versus Critical Care Patients
Brief Title: Evaluation of Oxidative Stress Induced by Iron Injection in Healthy Volunteers and Critical Care Patients
Acronym: SOFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P101104; 2011-000819-10 (EudraCT Number)
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Critical Illness
Keywords: iron; critical illness; oxidative stress
MeSH Terms: conditions — Critical Illness | interventions — Iron; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- critical care patients venofer (Experimental): Critically ill patients are injected with Venofer (ferric hydroxide sucrose) 100mg IV in one hour (in critically ill patients the injection could be repeated on day 2 (200mg) and 4 (100mg) depending on treatment
  Interventions: Drug: critical care patients venofer

INTERVENTIONS:
Drug: critical care patients venofer — 100mg IV in one hour (in critically ill patients the injection could be repeated on day 2 (200mg) and 4 (100mg) depending on treatment
  Other Names: iron (ferric hydroxide sucrose) injection

SUMMARY:
The purpose of this study is to evaluate the pro-oxidant toxicity of iron injections in critically ill patients and in healthy volunteers. The investigators hypothesize that the inflammatory state of critically ill patients will reduce the oxydative stress induced by iron injections, compared to the one induced in healthy volunteers. It will be an open "proof-of-concept" study aimed at evaluating iron toxicity in critically ill patients (n=40) as compared to healthy volunteers (n=40).

The investigators will compare the oxidative stress (principal judgment criteria= 8-iso-PGF2α) following a 100 mg injection of iron (at T0, T2, T6 and T24 hours post injection) in both groups and the investigators will compare the effect of repeated injections in the critically ill patients.

DETAILED DESCRIPTION:
Anemia is frequent among critically ill patients, with 60% of the patients being anemic at admission and more than 80% at discharge. This anemia is associated with an increased MORBI-mORTALITY. However, therapeutic options, mainly transfusion and erythropoietin, are disappointing. There is a remaining therapeutic option, iron injection, which has not been fully evaluated because of potential restrictions: inflammation may prevent its efficacy, and iron could be toxic, notably through the generation of oxidative stress. Our research is aimed at exploring the benefit of iron treatment in the critical care anemia.

The investigators already demonstrated in a MURIN model of critical care anemia that the master regulator of iron metabolism, hepcidin, is repressed and that iron can be mobilized from the stores despite inflammation. In addition, in an observational human study, the investigators reported that 25% of critically ill patients had iron deficiency and low to normal hepcidin levels.

All together, these data indicate that iron therapy may be beneficial in this situation. In the present study, the investigators evaluate the toxicity of iron in that context of critical care anemia. Iron, especially non-transferrin bound iron, is known to induce the generation of oxygen-derived free radicals through the Fenton reaction. However, the generation of oxidative stress secondary to iron injection has not been investigated in the critically ill. In our animal model, preliminary data indicate that the production of oxidative stress in the serum following iron injection may be prevented by inflammation.

Objectives: To evaluate the pro-oxidant toxicity of iron injections in critically ill patients and in healthy volunteers. The investigators hypothesize that the oxidative stress will be reduced in critically ill as compared to healthy volunteers

Human study : It will be an open "proof-of-concept" study aiming at evaluating iron toxicity in critically ill patients (n=40) as compared to healthy volunteers (n=40).

The investigators will compare the oxidative stress (principal judgment criteria= 8-iso-PGF2α) following a 100 mg injection of iron (at T0, T2, T6 and T24 hours post injection) in both groups and the investigators will compare the effect of repeated injections in the critically ill patients.

Perspectives:

This study should confirm that iron does not produce more oxidant stress in critically ill patients than in healthy volunteers. The animal study should help to precise the efficacy of this treatment, in addition to its toxicity. All these results will help to design a phase III randomized study of intravenous iron in critically ill anemic patients

ELIGIBILITY:
INCLUSION CRITERIA:

* Man or woman hospitalized in critical care unit,
* between 18 and 90 years old
* clinical examination completed
* written consent from the patient or a patient's relative depending on the awareness of the patient
* an iron injection has been prescribed by the responsible physician to the patient
* anemia defined as hemoglobin level ≤11 g/dl
* iron deficiency define by at least one of the following criteria :

  * ferritin < 100 μg/l
  * ferritin between 100 and 300 μg/l with transferrin saturation < 20%,
  * soluble transferrin receptor (RsTf) ≥1,4 mg/l,
  * ratio RsTf/log(ferritin) ≥0,7,
  * blood loss ≥ 1 blood weight.

EXCLUSION CRITERIA:

* do not subscribe to the french health insurance program
* Pregnancy or nursing
* past medical history of iron overload or disfunction in iron metabolism (= primary or secondary hemochromatosis)
* Recent bacteremia defined as positive in the 48 hours preceding the injection. Having a non positive hemoculture is not an exclusion criteria
* Suspicion of a novel current infection defined by a new fever with temperature over >38°5 for at least three times during the last 48hours. A persisting fever for more than 48 hours without argument for a new infection is not an exclusion criteria.
* known allergia to the iron- hydroxide complex or one of the excipient
* active chronic alcoholism
* oral iron treatment during the last 24 hours. Usage of antioxidant (vitamin C, vitamin E) within the 24 hours preceding the iron injection.
* person participating to another clinical trial or being in the exclusion phase of a clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
serum 8-iso-PGF2α | 0 hours
  oxidative stress
serum 8-iso-PGF2α | 2 hours
  oxidative stress
serum 8-iso-PGF2α | 6 hours
  oxidative stress
serum 8-iso-PGF2α | 24 hours
  oxidative stress

SECONDARY OUTCOMES:
Advanced Oxidized Protein Product | 0 hours
  oxidative stress
Advanced Oxidized Protein Product | 2 hours
  oxidative stress
Advanced Oxidized Protein Product | 6 hours
  oxidative stress
Advanced Oxidized Protein Product | 24 hours
  oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond Lasocki, MD PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Bichat-Claude Bernard, Paris, France